CLINICAL TRIAL: NCT00652275
Title: Phase IIb Immunogenicity, Efficacy and Safety Study of P. Falciparum Vaccine Candidate, MSP3-LSP Adjuvanted in Aluminium Hydroxide Versus Verorab Control in Healthy Children Aged 12-48 Months in Mali.
Brief Title: Immunogenicity, Efficacy and Safety Study of an MSP3-LSP (Long Synthetic Peptide) Malaria Vaccine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: African Malaria Network Trust (Network)
Responsible Party: Roma Chilengi, African Malaria Network Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MSP3_ML_0304; MMVDU-007
Record Dates: First submitted 2008-03-18; First posted 2008-04-03 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-04

CONDITIONS: Malaria
Keywords: Malaria; vaccine; Merozoite surface Antigene; Mali; Children
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Biological/Vaccine: 189 volunteers will receive the Malaria vaccine MSP3 Long Synthetic Peptide (LSP)
  Arms: MSP3 LSP vaccine Biological/Vaccine:MSP3 LSP 30 micrograms of MSP3 LSP
  Arms: I, MSP3 LSP vaccine
  Interventions: Biological: MSP3 Long Synthetic Peptide 30 micrograms of MSP3 LSP
- B (Active Comparator): 189 volunteers will receive standard vaccine against rabies on the similar schedule on days 0, 28, and 56
  Interventions: Biological: Verorab vaccine

INTERVENTIONS:
Biological: MSP3 Long Synthetic Peptide 30 micrograms of MSP3 LSP — 189 children will receive 3 doses of experimental vaccine
  Arms: A
Biological: Verorab vaccine — 189 volunteers will receive Verorab vaccine, 0.5 Ml at day 0, 28 and 56.
  Arms: B

SUMMARY:
This study will be the fourth time that the candidate malaria vaccine Merozoite Surface Protein - long synthetic chain, will be tested in malaria endemic populations.in the past,once tested in adults and twice in children proved to be safe in all three occasions for this phase IIb study in children to proceed. This study will include children who will be randomly allocated to either receive the malaria vaccine adjuvanted with Aluminium Hydroxide or the Verorab control. Each participant will receive 3 immunizations, without the clinical investigators or the participants themselves knowing what has been given. They will then be followed-up for immediate reactions to vaccination, extended safety profile and immunological response associated with protection from malaria. These children will be followed up for over a longer term of two years. Blood will be taken to evaluate the biological safety parameters and also the immune responses.

DETAILED DESCRIPTION:
This will be a double blind, randomized, placebo-controlled phase IIb study to evaluate the immunogenicity, efficacy and safety of Plasmodium falciparum vaccine candidate, Merozoite Surface Protein-3 Long synthetic peptide (MSP3) adjuvanted in aluminium hydroxide versus Verorab control in healthy children aged 12-48 months in Mali

A phase Ib trial is currently ongoing in Burkina Faso as well as in Tanzania and its interim results inform on the best dose/adjuvant combination to be safely extended in younger children. The trial is evaluating immunogenicity,efficacy and safety of 3 doses of 30 µg MSP3 adjuvanted in aluminium hydroxide

Primary objective:

* To assess the efficacy of MSP3-LSP:
* Determine the efficacy of MSP3-LSP in children aged 12-48 months against all clinical malaria episodes (Axillary temperature of ≥ 37.5ºC with P. falciparum parasitemia) occurring during the consecutive malaria transmission season after the third vaccination (six months after the third vaccination).

Secondary Objectives:

* To assess the safety and reactogenicity of 3 doses of 30 µg MSP3 adjuvanted in aluminum hydroxide given at D0, D28 and D56 in healthy children aged 12-48 months old in Mali.
* To assess IgG ability to recognize the native protein on Merozoite by using Western Blot (WB) method, and measure efficacy among the subgroup of individuals able to react with parasite proteins in WB.
* To assess the humoral immune response to the vaccine antigen using ELISA.
* Determine the efficacy of MSP3 in children aged 12-48 months against first clinical malaria episodes.
* To assess the efficacy of MSP3-LSP in children aged 12-48 months against all clinical malaria episodes occurring during the ensuing TWO years

Exploratory Objectives:

To further characterize the MSP3 vaccine efficacy by measuring:

* Relationship between efficacy and serological responses induced by the vaccine
* Duration of protection over the period of two years
* Vaccine efficacy against disease defined by various parasite thresholds [500, 2500, 5000, 10,000 and 20,000/µL]
* Vaccine efficacy against severe malaria disease
* Vaccine efficacy against anaemia
* To evaluate functionality of IgG by using the ADCI technique
* To assess the cellular T-helper type 1 immune responses to the vaccine antigens by Elispot, and their persistence over 24 months of follow-up

The primary evaluation will include the following:

Solicited adverse events measured from day 0 to day 7 after each dose; Unsolicited adverse events measured up to one month after each dose; Serious Adverse Event (SAE) measured during the 12 months of study duration. Passive and active case detection will be used to capture all adverse events including clinical malaria episodes. After third dose. All participants will go through the scheduled clinic visits on days 84, 168, 365, 540 and 730 for clinical assessment. Children will be followed for two years following the first vaccination. During scheduled visits malaria smear and hemoglobin will be done systematically on days 0, 28, 56, 84, 168, 365, 540 and 730. The humoral immune response to the vaccine antigen will be assessed using ELISA on days 0, 28, 56, 84, 168, 365, 540 and 730. Cellular immune response to the vaccine antigens will be assessed on days 0, 56, 84, 168, 540 and 730 using Elispot to MSP3-LSP. The functionality of the induced immune responses using Western Blot (WB) method and ADCI technique will be evaluated on days 0, 84, 168, 365, 540 and 730.

Biological safety: two and four weeks after each vaccination, and thereafter every 12 weeks, in reference with the baseline before the first dose, by measuring the following RBC, hemoglobin, hematocrit, platelets, WBC with differential counts, ASAT, ALAT, total bilirubin, alkaline phosphatase, γGT, creatinin.

Statistical methods:

Descriptive methods shall be employed to evaluate the above criteria.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 12-48 months old
* Healthy by medical history, physical examination and laboratory investigation
* Signed/thumb printed informed Consent by guardian/parent
* Resident in the study area villages during the whole trial period

Exclusion Criteria:

* Symptoms, physical signs of disease that could interfere with the interpretation of the trial results or compromising the health of the subjects
* Immunosuppressive therapy (steroids, immune modulators or immune suppressors) within 3 months prior recruitment. (Inhaled and topical steroids are allowed).
* Cannot be followed for any social, psychological or geographical reasons.
* Use of any investigational drug or vaccine other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use up to 30 days after the third dose.
* Suspected or known hypersensitivity to any of the vaccine components or to previous vaccine.
* Laboratory abnormalities on screened blood samples.
* Planned administration of a vaccine not foreseen by the study protocol within 30 days before the first dose of vaccine. An exception, is the receipt of an EPI or licensed vaccine (measles, oral polio, Hib, meningococcal and combined diphtheria/pertussis/tetanus vaccines) which may be given 14 days or more before or after vaccination
* Evidence of chronic or active hepatitis B or C infection
* Presence of chronic illness that, in the judgment of the investigator, would interfere with the study outcomes or pose a threat to the participant's health.
* Administration of immunoglobulin and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period
* History of surgical splenectomy.
* Moderate or severe malnutrition at screening defined as weight for age Z-score less than 2

Ages: 12 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 378 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-11 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Number of clinical malaria episodes occurring during the consecutive malaria transmission season after the third vaccination | 27 Months

SECONDARY OUTCOMES:
Solicited adverse events measured from day 0 to day 7 after each dose | 7 days
Unsolicited adverse events measured up to one month after each dose | Day 84
Serious Adverse Events measured during the 12 months of study duration | 2 years
The humoral response to the vaccine antigen: assessed by measuring the level of IgG by ELISA | Day 84
IgG ability to recognize the native protein on Merozoite using Western Blot(WB) method | Day 84
Incidence of all clinical malaria episodes occurring through two transmission seasons subsequent to the 3 doses. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mahamadou S Sissoko, MD, MSPH, Principal Investigator — Malaria Research and Training Center (MRTC), Bamako Mali; Roma Chilengi, MBChB, MSc, Study Director — African Malaria Network Trust
Locations (1):
- Malaria Research Training Center, Bamako, Mali